CLINICAL TRIAL: NCT01937949
Title: Clinical Outcomes and Quality of Life Measures in Patients Treated for Complex Abdominal Aortic Aneurysms With Fenestrated Stent Grafts
Brief Title: Complex Abdominal Aortic Aneurysm Repair With Fenestrated Stent Grafts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustavo S Oderich (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Gustavo S Oderich, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-57286
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Juxtarenal Aortic Aneurysms; Suprarenal Aortic Aneurysms; Type IV Thoracoabdominal Aortic Aneurysms
Keywords: Aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endovascular (Other): The study will include patients treated by endovascular aortic repair of juxtarenal, suprarenal and type IV thoracoabdominal aortic aneurysms using custom-made Cook Zenith® Fenestrated AAA Endovascular Graft. The graft includes combinations of scallops, holes (fenestrations) or cuffs (side branches) . These small holes or branches are the investigational part of this research study. The arteries to the liver, intestine, and kidneys will be have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches.
  Other names:
  Endovascular stent Stent-graft
  Interventions: Device: Custom-made Zenith® Fenestrated AAA Endovascular Graft:

INTERVENTIONS:
Device: Custom-made Zenith® Fenestrated AAA Endovascular Graft: — The graft will be inserted through arteries in the groin (called endovascular repair). Endovascular repair is a procedure that uses catheters that go inside your blood vessel to place a stent graft above and below the aneurysm. This procedure lines the aneurysm with a new lining (stent) so blood does not fill the artery any more.
  Other Names: Endovascular stent; Stent-graft

SUMMARY:
The purpose of this study is to evaluate clinical outcomes and quality of life measures in treated by endovascular aortic repair of juxtarenal, suprarenal, and type IV thoracoabdominal aortic aneurysms using custom-made Cook Zenith® Fenestrated AAA Endovascular Graft.

DETAILED DESCRIPTION:
This is a traditional device feasibility study intended to generate preliminary safety and efficacy information that may be used to plan an appropriate future study, or to inform further product development.

ELIGIBILITY:
General Inclusion Criteria

* A patient may be included in the study if the patient has at least one of the following and is appropriate for treatment with a custom-made Zenith® Fenestrated AAA Endovascular Graft:
* Juxtarenal, suprarenal or type IV thoracoabdominal aortic aneurysm with a diameter ≥ 5.0 cm or 2 times the normal aortic diameter
* Aneurysm with a history of growth ≥ 0.5 cm per year
* Saccular aneurysms deemed at significant risk for rupture based upon physician interpretation.

General Exclusion Criteria

* Less than 18 years of age
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Pregnant or breastfeeding
* Life expectancy < 2-years
* Additional medical restrictions as specified in the Clinical Investigation Plan
* Additional anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who have die at 30 days post treatment | 30 days post treatment]
  Deaths 30 days after treatment
Number of subjects who experience a Major Adverse Event at 30 days post treatment | 30 days post treatment
  A Major Adverse Event includes any of the following: bowel ischemia, myocardial infarction (heart attack), paraplegia, renal failure, respiratory failure, stroke, or blood loss greater than 1000 ml.

SECONDARY OUTCOMES:
Subject Scores on Short Form-36 (SF-36) Quality of Life Questionnaire | baseline, 6 weeks, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years.
  Subjects completed the SF-36 which consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
Number of Subjects Who Achieve Treatment Success | 12 months
  Treatment success is defined by a composite end-point, which includes all the following criteria described below:
  * Technical success, defined as successful delivery and deployment of the custom-made endovascular graft with preservation of those branch vessels intended to be preserved.
  * Freedom from type I or III endoleak.
  * Freedom from stent-graft migration.
  * Freedom from aneurysm enlargement >5mm
  * Freedom from aneurysm rupture or conversion to open repair.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo S. Oderich, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cirillo-Penn NC, MacArthur TA, Tenorio ER, DeMartino RR, Macedo TA, Oderich GS, Mendes BC. Outcomes of patients treated with double-wide scallop vs fenestrations for celiac artery incorporation during repair of complex abdominal aortic aneurysms. J Vasc Surg. 2025 May;81(5):1033-1039. doi: 10.1016/j.jvs.2025.01.194. Epub 2025 Jan 28. PMID 39884565
- [Result] Finnesgard EJ, Jones DW, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Schanzer A; United States Aortic Research Consortium. Trends and outcomes over time with fenestrated and branched endovascular aortic repair in the United States Aortic Research Consortium. J Vasc Surg. 2025 Jun;81(6):1235-1243. doi: 10.1016/j.jvs.2025.01.213. Epub 2025 Feb 4. PMID 39914755
- [Result] Vacirca A, Mesnard T, Huang Y, Mendes BC, Jakimowicz T, Schneider DB, Haulon S, Sobocinski J, Beck AW, Schanzer A, Farber MA, Timaran C, Kahlberg A, Kolbel T, Gasper WJ, Mees BME, Gargiulo M, Dias NV, Woongchae AL, Sweet MP, Mani K, Eagleton M, Pedro LM, Verhagen H, Yeung KK, Tsilimparis N, Resch T, Bertoglio L, Ferreira E, Khashram M, Sulzer T, Dias-Neto M, Tenorio ER, Kanamori LR, Jama K, Parodi E, Gomes V, Colon JP, Chiesa R, Panuccio G, Schurink GW, Lemmens C, Gallitto E, Faggioli G, Karelis A, Wanhainen A, Habib M, Gouveia E Melo R, Kappe KO, Mariko van Knippenberg SE, Tran B, Crawford S, Panagrosso M, Melloni A, Bonardelli S, Garcia R, Ribeiro T, Gormley S, Maximus S, Oderich GS; International Multicenter Aortic Research Group. Predictors of failure to rescue after fenestrated-branched endovascular aortic repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2025 Jul;82(1):32-42.e3. doi: 10.1016/j.jvs.2025.02.032. Epub 2025 Mar 5. PMID 40054790
- [Result] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Result] Ruiter Kanamori L, Tenorio E, Babocs D, Lima GB, Mendes B, Macedo TA, Maximus S, Huang Y, Oderich GS. Clinical outcomes and quality of life measures among 5-year survivors of fenestrated-branched endovascular aortic repair. J Vasc Surg. 2025 Jun;81(6):1254-1265. doi: 10.1016/j.jvs.2025.01.210. Epub 2025 Feb 2. PMID 39904414
- [Result] Chait J, Tenorio ER, Kawajiri H, Lima GBB, Cirillo-Penn NC, Bagameri G, Pochettino A, DeMartino RR, Oderich GS, Mendes BC. Mid-Term Outcomes of "Complete Aortic Repair": Surgical or Endovascular Total Arch Replacement With Thoracoabdominal Fenestrated-Branched Endovascular Aortic Repair. J Endovasc Ther. 2025 Apr;32(2):503-512. doi: 10.1177/15266028231181211. Epub 2023 Jun 14. PMID 37313951
- [Result] Ruiter Kanamori L, Tenorio ER, Babocs D, Savadi S, Baghbani-Oskouei A, Huang Y, Figueroa A, Tanenbaum M, Costa Filho JE, Baig M, Macedo TA, Timaran CH, Oderich GS. Indications, safety, and effectiveness of transcatheter electrosurgical septotomy during endovascular repair of aortic dissections. J Vasc Surg. 2024 Nov;80(5):1396-1406. doi: 10.1016/j.jvs.2024.07.089. Epub 2024 Jul 27. PMID 39074740
- [Result] Huang Y, Colglazier J, Mendes BC, Pochettino A, Kalra M, Greason KL, Tenorio ER, Harmsen WS, Oderich GS. Target Artery Outcomes Following Endovascular versus Open Surgical Repair of Thoracoabdominal Aortic Aneurysms - A Single Center Comparative Study. Ann Surg. 2024 Nov 25. doi: 10.1097/SLA.0000000000006594. Online ahead of print. PMID 39584778
- [Result] Steadman JA, Tenorio ER, Chait J, Vierkant RA, DeMartino RR, Oderich GS, Mendes BC. Preoperative predictors of nonhome discharge after fenestrated-branched endovascular repair of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2024 Mar;79(3):469-477.e3. doi: 10.1016/j.jvs.2023.11.015. Epub 2023 Nov 11. PMID 37956958
- [Result] Mesnard T, Vacirca A, Baghbani-Oskouei A, Sulzer TAL, Savadi S, Kanamori LR, Tenorio ER, Mirza A, Saqib N, Mendes BC, Huang Y, Oderich GS. Prospective evaluation of upper extremity access and total transfemoral approach during fenestrated and branched endovascular repair. J Vasc Surg. 2024 May;79(5):1013-1023.e3. doi: 10.1016/j.jvs.2023.12.033. Epub 2023 Dec 21. PMID 38141739
- [Result] Blakeslee-Carter J, Novak Z, Jansen JO, Schanzer A, Eagleton MJ, Farber MA, Gasper W, Lee WA, Oderich GS, Timaran CH, Schneider DB, Sweet MP, Beck AW. Prospective randomized pilot trial comparing prophylactic and therapeutic cerebrospinal fluid drainage during complex endovascular thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2024 Jul;80(1):11-19. doi: 10.1016/j.jvs.2024.02.041. Epub 2024 Apr 6. PMID 38614137
- [Result] Tanenbaum MT, Figueroa AV, Kanamori LR, Costa Filho JE, Soto Gonzalez M, Sulzer T, Mesnard T, Huang Y, Baig MS, Oderich GS, Timaran CH. Early experience with patient-specific unibody bifurcated fenestrated-branched devices for complex endovascular aortic aneurysm repair. J Vasc Surg. 2024 Nov;80(5):1361-1370. doi: 10.1016/j.jvs.2024.06.020. Epub 2024 Jun 17. PMID 38897392
- [Result] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Result] Tenorio ER, Mirza AK, Lima GBB, Marcondes GB, Wong J, Mendes BC, Saqib N, Khan S, Macedo TA, Oderich GS. Characterization of Secondary Interventions After Fenestrated-branched Endovascular Repair of Complex Aortic Aneurysms and Its Effect on Quality of Life and Patient Survival. Ann Surg. 2023 Jul 1;278(1):140-147. doi: 10.1097/SLA.0000000000005454. Epub 2022 Jul 8. PMID 35801701
- [Result] Dias-Neto M, Marcondes G, Tenorio ER, Barbosa Lima GB, Baghbani-Oskouei A, Vacirca A, Mendes BC, Saqib N, Mirza AK, Oderich GS. Outcomes of iliofemoral conduits during fenestrated-branched endovascular repair of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Mar;77(3):712-721.e1. doi: 10.1016/j.jvs.2022.10.050. Epub 2022 Nov 5. PMID 36343871
- [Result] Vacirca A, Wong J, Baghbani-Oskouei A, Tenorio ER, Huang Y, Mirza A, Saqib N, Sulzer T, Mesnard T, Mendes BC, Oderich GS. Outcomes of fenestrated-branched endovascular aortic repair in patients with or without prior history of abdominal endovascular or open surgical repair. J Vasc Surg. 2023 Aug;78(2):278-288.e3. doi: 10.1016/j.jvs.2023.04.001. Epub 2023 Apr 19. PMID 37080442
- [Result] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Result] Paajanen P, Karkkainen JM, Tenorio ER, Mendes BC, Oderich GS. Effect of patient frailty status on outcomes of fenestrated-branched endovascular aortic repair for complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2022 Nov;76(5):1170-1179.e2. doi: 10.1016/j.jvs.2022.05.008. Epub 2022 Jun 11. PMID 35697310
- [Result] Dias-Neto M, Tenorio ER, Lima GBB, Baghbani-Oskouei A, Saqib N, Mendes BC, Mirza AK, Oderich GS. Outcomes of low- and standard-profile fenestrated and branched stent grafts for treatment of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2022 Nov;76(5):1160-1169.e1. doi: 10.1016/j.jvs.2022.05.028. Epub 2022 Jul 8. PMID 35810953
- [Result] Chait J, Tenorio ER, Mendes BC, Barbosa Lima GB, Marcondes GB, Wong J, Macedo TA, De Martino RR, Oderich GS. Impact of gap distance between fenestration and aortic wall on target artery instability following fenestrated-branched endovascular aortic repair. J Vasc Surg. 2022 Jul;76(1):79-87.e4. doi: 10.1016/j.jvs.2022.01.135. Epub 2022 Feb 16. PMID 35181519
- [Result] Tenorio ER, Ribeiro MS, Banga PV, Mendes BC, Karkkainen J, DeMartino RR, Hoffman EM, Oderich GS. Prospective Assessment of a Protocol Using Neuromonitoring, Early Limb Reperfusion, and Selective Temporary Aneurysm Sac Perfusion to Prevent Spinal Cord Injury During Fenestrated-branched Endovascular Aortic Repair. Ann Surg. 2022 Dec 1;276(6):e1028-e1034. doi: 10.1097/SLA.0000000000004624. Epub 2021 Jan 7. PMID 33417331
- [Result] Squizzato F, Oderich GS, Tenorio ER, Mendes BC, DeMartino RR. Effect of celiac axis compression on target vessel-related outcomes during fenestrated-branched endovascular aortic repair. J Vasc Surg. 2021 Apr;73(4):1167-1177.e1. doi: 10.1016/j.jvs.2020.07.092. Epub 2020 Aug 27. PMID 32861863
- [Result] Squizzato F, Oderich GS, Balachandran P, Tenorio ER, Mendes BC, De Martino RR. Effect of aortic angulation on the outcomes of fenestrated-branched endovascular aortic repair. J Vasc Surg. 2021 Aug;74(2):372-382.e3. doi: 10.1016/j.jvs.2021.01.027. Epub 2021 Feb 4. PMID 33548434
- [Result] Karkkainen JM, Oderich GS, Tenorio ER, Pather K, Oksala N, Macedo TA, Vrtiska T, Mees B, Jacobs MJ. Psoas muscle area and attenuation are highly predictive of complications and mortality after complex endovascular aortic repair. J Vasc Surg. 2021 Apr;73(4):1178-1188.e1. doi: 10.1016/j.jvs.2020.08.141. Epub 2020 Sep 28. PMID 33002587
- [Result] Marcondes GB, Tenorio ER, Baumgardt G, Mendes B, Oderich GS. Evaluation of Safety of Overhead Upper Extremity Positioning During Fenestrated-Branched Endovascular Repair of Thoracoabdominal Aortic Aneurysms. Cardiovasc Intervent Radiol. 2021 Dec;44(12):1895-1902. doi: 10.1007/s00270-021-02992-1. Epub 2021 Oct 27. PMID 34708266
- [Result] Banga P, Oderich GS, Farber M, Reis de Souza L, Tenorio ER, Timaran C, Schneider DB, Baumgardt Barbosa Lima G, Barreira Marcondes G, Timaran D. Impact of Number of Vessels Targeted on Outcomes of Fenestrated-Branched Endovascular Repair for Complex Abdominal Aortic Aneurysms. Ann Vasc Surg. 2021 Apr;72:98-105. doi: 10.1016/j.avsg.2020.09.063. Epub 2020 Nov 21. PMID 33227467
- [Result] Oderich GS, Tenorio ER, Mendes BC, Lima GBB, Marcondes GB, Saqib N, Hofer J, Wong J, Macedo TA. Midterm Outcomes of a Prospective, Nonrandomized Study to Evaluate Endovascular Repair of Complex Aortic Aneurysms Using Fenestrated-Branched Endografts. Ann Surg. 2021 Sep 1;274(3):491-499. doi: 10.1097/SLA.0000000000004982. PMID 34132698
- [Result] Sen I, Tenorio ER, Mirza AK, Karkkainen JM, Mendes BC, DeMartino RR, Cha S, Oderich GS. Effect of Blood Loss and Transfusion Requirements on Clinical Outcomes of Fenestrated-Branched Endovascular Aortic Repair. Cardiovasc Intervent Radiol. 2020 Nov;43(11):1600-1607. doi: 10.1007/s00270-020-02573-8. Epub 2020 Aug 30. PMID 32864718
- [Result] Karkkainen JM, Tenorio ER, Pather K, Mendes BC, Macedo TA, Wigham J, Diderrich A, Oderich GS. Outcomes of Small Renal Artery Targets in Patients Treated by Fenestrated-Branched Endovascular Aortic Repair. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):910-917. doi: 10.1016/j.ejvs.2020.02.015. Epub 2020 Mar 18. PMID 32197996
- [Result] Karkkainen JM, Tenorio ER, Jain A, Mendes BC, Macedo TA, Pather K, Gloviczki P, Oderich GS. Outcomes of target vessel endoleaks after fenestrated-branched endovascular aortic repair. J Vasc Surg. 2020 Aug;72(2):445-455. doi: 10.1016/j.jvs.2019.09.055. Epub 2020 Jan 21. PMID 31980247
- [Result] Tenorio ER, Karkkainen JM, Mendes BC, DeMartino RR, Macedo TA, Diderrich A, Hofer J, Oderich GS. Outcomes of directional branches using self-expandable or balloon-expandable stent grafts during endovascular repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2020 May;71(5):1489-1502.e6. doi: 10.1016/j.jvs.2019.07.079. Epub 2019 Oct 11. PMID 31611106
- [Result] Chini J, Mendes BC, Tenorio ER, Ribeiro MS, Sandri GA, Cha S, Hofer J, Oderich GS. Preloaded Catheters and Guide-Wire Systems to Facilitate Catheterization During Fenestrated and Branched Endovascular Aortic Repair. Cardiovasc Intervent Radiol. 2019 Dec;42(12):1678-1686. doi: 10.1007/s00270-019-02322-6. Epub 2019 Aug 27. PMID 31455986
- [Result] Karkkainen JM, Sandri GA, Tenorio ER, Macedo TA, Hofer J, Gloviczki P, Cha S, Oderich GS. Prospective assessment of health-related quality of life after endovascular repair of pararenal and thoracoabdominal aortic aneurysms using fenestrated-branched endografts. J Vasc Surg. 2019 May;69(5):1356-1366.e6. doi: 10.1016/j.jvs.2018.07.060. Epub 2018 Oct 24. PMID 30714570
- [Result] Oderich GS, Ribeiro M, Reis de Souza L, Hofer J, Wigham J, Cha S. Endovascular repair of thoracoabdominal aortic aneurysms using fenestrated and branched endografts. J Thorac Cardiovasc Surg. 2017 Feb;153(2):S32-S41.e7. doi: 10.1016/j.jtcvs.2016.10.008. Epub 2016 Oct 22. PMID 27866781
- [Result] Oderich GS, Ribeiro M, Hofer J, Wigham J, Cha S, Chini J, Macedo TA, Gloviczki P. Prospective, nonrandomized study to evaluate endovascular repair of pararenal and thoracoabdominal aortic aneurysms using fenestrated-branched endografts based on supraceliac sealing zones. J Vasc Surg. 2017 May;65(5):1249-1259.e10. doi: 10.1016/j.jvs.2016.09.038. Epub 2016 Dec 13. PMID 27986479
- [Result] Banga PV, Oderich GS, Reis de Souza L, Hofer J, Cazares Gonzalez ML, Pulido JN, Cha S, Gloviczki P. Neuromonitoring, Cerebrospinal Fluid Drainage, and Selective Use of Iliofemoral Conduits to Minimize Risk of Spinal Cord Injury During Complex Endovascular Aortic Repair. J Endovasc Ther. 2016 Feb;23(1):139-49. doi: 10.1177/1526602815620898. Epub 2015 Dec 4. PMID 26637837
- [Result] Jain V, Banga P, Vallabhaneni R, Eagleton M, Oderich G, Farber MA. Endovascular treatment of aneurysms using fenestrated-branched endografts with distal inverted iliac limbs. J Vasc Surg. 2016 Sep;64(3):600-4. doi: 10.1016/j.jvs.2016.02.058. PMID 27565586